CLINICAL TRIAL: NCT05970328
Title: HMS ECG Clinical Validation Study - Protocol External Site
Brief Title: Hexoskin Medical System - ECG Performance Testing
Status: Completed | Type: Observational
Sponsor: Carré Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HMSECG23; 361070 (Other: Health Canada Investigation Testing Authorization)
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Rhythm Disturbance
Keywords: Hexoskin Medical System (HMS); Cardiac Rhythm Disturbance
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arrhythmia Participant: Non-critical adult (21 years and older) participants that are suspected of having an arrhythmia or have evidence of arrhythmia requiring monitoring via 24-hour Holter monitor.
  Interventions: Device: Hexoskin Medical System

INTERVENTIONS:
Device: Hexoskin Medical System — Participant wears both the Hexoskin Medical System and the Nasiff Holter Monitor at the same time to acquire ECG recordings.
  Other Names: Nasiff Holter Monitor

SUMMARY:
The goal of this observational study is to validate the efficacy of the Hexoskin Medical System (HMS) for its intended use (i.e., manual assessment of cardiac rhythm disturbances) in non-critical adult participants who are suspected of having an arrhythmia or have evidence of arrhythmia requiring monitoring via 24-hour Holter monitor.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

1. Whether the HMS ECG recordings can be used to accurately detect cardiac beats when compared with the Holter monitor
2. Whether there are good agreements between the HMS and Holter monitor in ECG characteristics
3. Whether the HMS ECG recordings can be used to accurately classify cardiac rhythm/rhythm disturbance when compared with the Holter monitor
4. What is the accuracy of using HMS ECG recordings to detect cardiac beats
5. What is the accuracy of using HMS ECG recordings to identify cardiac rhythm/rhythm disturbance

Participants will wear the HMS and the Holter monitor at the same time to record ECG signals. Researchers will evaluate the ECG recordings acquired from both devices and assess the above questions.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 21 years or older.
* Participants must be suspected of having an arrhythmia or have evidence of arrhythmia requiring monitoring via 24-hour Holter monitor.

Exclusion Criteria:

* Body circumference that is not covered by the HMS Shirt sizing chart
* Presence of pacemaker or Implantable Cardioverter-Defibrillator (ICD) devices
* Known allergic reactions to silver or polyamide/polyester/elastane
* Known allergic reactions to ECG gel electrodes
* Documented medical condition or illness requiring intensive medical treatment or care

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients consulting the cardiology clinics
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
ECG characteristics measurement agreement | 2 days
  The agreement (Bland-Altman plots) of Holter monitor(reference standard) and HMS to measure each of the four (4) ECG Characteristics. ECG characteristics measured in this study include: RR Interval (ms), PR Interval (ms), PP Interval (ms), and QRS Duration (ms).

SECONDARY OUTCOMES:
Heart rate agreement | 2 days
  The agreement between HR calculated from the recordings acquired by the subject device and the reference Holter monitor.

OTHER OUTCOMES:
Cardiac beat detection accuracy | 2 days
  The sensitivity and PPV of using the subject device recordings to detect cardiac beats.
Rhythm identification accuracy | 2 days
  The sensitivity and PPV of using the subject recordings to identify cardiac rhythm/rhythm disturbances.
ECG recording stability | 2 days
  The stability of the subject device for recording ECG through 24 hours of ambulatory ECG monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cheung, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Lawrence Park Cardiology, Toronto, Ontario
  - Yorkview Cardiology, North York

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.